CLINICAL TRIAL: NCT05986032
Title: Relationship Between Respiratory System Reactance Assessed by Respiratory Oscillometry and Respiratory Outcomes in Very Preterm Infants
Brief Title: Respiratory Oscillometry for the Prediction of Bronchopulmonary Dysplasia
Acronym: REACT
Status: Recruiting | Type: Observational
Sponsor: Fondazione IRCCS San Gerardo dei Tintori (Other)
Collaborators: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other); University Children's Hospital Basel (Other); Uppsala University Hospital (Other); Medical University of Vienna (Other); Amsterdam University Medical Centers (UMC), Location Academic Medical Center (AMC) (Other)
Responsible Party: Sponsor
Other Study IDs: REACT
Record Dates: First submitted 2023-07-19; First posted 2023-08-14 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Bronchopulmonary Dysplasia
Keywords: Respiratory oscillometry; Respiratory system reactance; Lung mechanics; Infant lung function testing
MeSH Terms: conditions — Bronchopulmonary Dysplasia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- no bronchopulmonary dysplasia: Group of patients who do not receive the diagnosis of bronchopulmonary dysplasia defined as the need for respiratory support at 36 weeks post-mentrual age
  Interventions: Diagnostic Test: Respiratory Oscillometry
- bronchopulmonary dysplasia: Group of patients developing bronchopulmonary dysplasia defined as the need for respiratory support at 36 weeks post-menstrual age.
  Interventions: Diagnostic Test: Respiratory Oscillometry

INTERVENTIONS:
Diagnostic Test: Respiratory Oscillometry — Measurement of respiratory system reactance by respiratory oscillometry

SUMMARY:
The goal of this observational study is to learn about the correlation between respiratory system reactance, as assessed by respiratory oscillometry, and respiratory outcomes in preterm infants born before 32 weeks of gestation. The main question it aims to answer is if the reactance z-score at 7 postnatal days adds to relevant clinical factors in the prediction of bronchopulmonary dysplasia. Participants will receive respiratory oscillometry measurements at 7 ± 2 postnatal days.

ELIGIBILITY:
Inclusion Criteria:

* born before 32 weeks post-menstrual age

Exclusion Criteria:

* congenital abnormalities
* Inherited disorders of metabolism

Ages: 5 Days to 9 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infants will be recruited from those admitted to tertiary-level neonatal intensive care units.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-07-15 (Actual); Primary Completion 2024-09-03 (Estimated); Study Completion 2024-09-24 (Estimated)

PRIMARY OUTCOMES:
Respiratory system reactance (Xrs) at the clinical positive end-expiratory pressure | Xrs will be measured at 7 days of life
  Xrs will be expressed in z-score using reference equation for very preterm infants

SECONDARY OUTCOMES:
Respiratory system reactance (Xrs) at the clinical positive end-expiratory pressure and ± 2 cmH2O | Xrs will be measured at 7 days of life
  Xrs will be expressed in cmH2O*S/L

OTHER OUTCOMES:
Respiratory support mode | 7 postnatal days
  Respiratory support mode will be coded as 0 = no respiratory support, 1 = nasal high flow therapy, 2 = nasal CPAP or nasal IPPV, 3 = invasive mechanical ventilation
Fraction of inspired oxygen | 7 days of life

CONTACTS AND LOCATIONS:
Overall Officials: Camilla Rigotti, PhD, Principal Investigator — Fondazione IRCCS San Gerardo dei Tintori
Locations (6):
- Medical University of Vienna, Vienna, Vienna, Austria
- Italy (2):
  - Fondazione IRCCS San Gerardo dei Tintori, Monza, Monza E Brianza
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan
- Amsterdam UMC, Amsterdam, Netherlands
- Uppsala University Children's Hospital, Uppsala, Sweden
- Universitäts-Kinderspital beider Basel, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zannin E, Neumann RP, Dellaca R, Schulzke SM. Forced oscillation measurements in the first week of life and pulmonary outcome in very preterm infants on noninvasive respiratory support. Pediatr Res. 2019 Sep;86(3):382-388. doi: 10.1038/s41390-019-0432-6. Epub 2019 May 20. PMID 31108499
- [Background] Veneroni C, Wallstrom L, Sindelar R, Dellaca' RL. Oscillatory respiratory mechanics on the first day of life improves prediction of respiratory outcomes in extremely preterm newborns. Pediatr Res. 2019 Feb;85(3):312-317. doi: 10.1038/s41390-018-0133-6. Epub 2018 Aug 4. PMID 30127523